CLINICAL TRIAL: NCT04867213
Title: Breath Analysis of Patients Diagnosed With COVID-19 Using Infrared Spectroscopy
Acronym: BREATH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Collaborators: Breathe BioMedical Inc (Industry)
Responsible Party: Principal Investigator, MyLinh Duong, Professor Department of Medicine, McMaster University
Other Study IDs: 12815
Record Dates: First submitted 2021-04-24; First posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: SARS-CoV-2 Infection; Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SARS-CoV-2 Positive: Clinically tested for SARS-CoV-2 (as completed by standard laboratory testing e.g. RT-PCR) and with a positive result and clinical features in keeping with COVID-19 illness. The investigators aim to collect breath samples within 7 days of symptom onset in 50% of Covid positive patients, with the remaining patients breath samples collected after 7 days of symptoms onset.
- SARS-CoV-2 Negative: Patients with a negative RT-PCR COVID-19 test and without any clinical features to suggest COVID-19 illness.

SUMMARY:
To analyze Volatile Organic Compounds (VOCs) in the breath of patients with SARS-CoV-2 and controls in SARS-CoV-2 breath specimens.

DETAILED DESCRIPTION:
The study is a prospective cohort study, which enrol patients presenting to hospital and are tested for SARS-CoV-2. There will be two cohorts, COVID-19 positive and COVID-19 negative, who will have exhaled breath collection and analysis by infrared spectroscopy to characterize the composition of VOCs and identify differences in VOC profiles between the two groups.

ELIGIBILITY:
Inclusion Criteria for Covid-19 positive patients:

* Clinically tested for SARS-CoV-2 (as completed by standard laboratory testing e.g. RT-PCR) with a positive result
* Clinical features in keeping with COVID-19 illness.

Inclusion criteria for Covid-19 negative patients:

* Negative RT-PCR COVID-19 test
* Without any clinical features to suggest COVID-19 illness.
* No known or current features of respiratory infection, COPD, asthma, interstitial lung disease, other respiratory inflammatory conditions or lung cancer.
* Able to provide a breath sample (as based on clinical judgement).

Exclusion Criteria for Covid-19 positive and negative patients:

- Unable to provide a breath sample

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Breath VOCs in covid positive and negative patients. | Through study completion, an average of 1 year
  To examine Volatile Organic Compounds (VOCs) by infrared spectroscopy in the breath of patients with SARS-CoV-2 and controls to determine if VOCs within a breath sample can differentiate Covid-19 positive from Covid-19 negative patients.

SECONDARY OUTCOMES:
Effect of time of symptom onset on VOCs in Covid-19 positive patients | Through study completion, an average of 1 year
  To examine the effect of time of symptom onset on VOCs in the breath of Covid-19 positive patients. The investigators aim to collect breath samples within 7 days of symptom onset in 50% of Covid positive patients, with the remaining patients breath samples collected after 7 days of symptoms onset.

CONTACTS AND LOCATIONS:
Overall Officials: Mylinh Duong, MD, Principal Investigator — McMaster University Hospital
Locations (1):
- Hamilton Health Sciences, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Cusack RP, Larracy R, Morrell CB, Ranjbar M, Le Roux J, Whetstone CE, Boudreau M, Poitras PF, Srinathan T, Cheng E, Howie K, Obminski C, O'Shea T, Kruisselbrink RJ, Ho T, Scheme E, Graham S, Beydaghyan G, Gavreau GM, Duong M. Machine learning enabled detection of COVID-19 pneumonia using exhaled breath analysis: a proof-of-concept study. J Breath Res. 2024 Mar 13;18(2). doi: 10.1088/1752-7163/ad2b6e. PMID 38382095